CLINICAL TRIAL: NCT07025408
Title: A Multicentre, Randomised, Double-blind, Dose-exploratory, Controlled Drug and Placebo-controlled Phase II Clinical Trial Evaluating the Safety, Efficacy, Pharmacokinetic Profile, and Immunogenicity of KJ101 for Wound Debridement in Deep II Degree Burns
Brief Title: Phase II Clinical Trial of KJ101in the Treatment of Deep II Degree Burns
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Bao Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHBJ-KJ101-002
Record Dates: First submitted 2025-06-10; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Burn; Burn Wounds - Partial Thickness (2nd Degree)
MeSH Terms: conditions — Burns | interventions — Chymotrypsin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental-KJ101-Dose Group -1 (Experimental): KJ101 , Dose Group -1 (800 U/mL)
  Interventions: Drug: KJ101
- Experimental-KJ101-Dose Group -2 (Experimental): KJ101 , Dose Group -2 (1200 U/mL)
  Interventions: Drug: KJ101
- Active comparator (Active Comparator): Chymotrypsin (800 U/mL)
  Interventions: Drug: Chymotrypsin
- Placebo Comparator (Placebo Comparator): Placebo
  Interventions: Drug: Placebo (Sodium Chloride Injection 0.9%)

INTERVENTIONS:
Drug: KJ101 — 1. Clean the wound before applying medication.
  2. Apply KJ101 (800U/mL) to the wound.
  3. Apply a standard wound dressing after treatment.
  4. Apply once daily until complete debridement of necrotic tissue has been achieved. After debridement, apply the medication every other day until the wound closes (maximum treatment duration: 28 days).
  Arms: Experimental-KJ101-Dose Group -1; Experimental-KJ101-Dose Group -2
Drug: Chymotrypsin — 1. Clean the wound before applying medication.
  2. Apply Chymotrypsin (800U/mL) to the wound.
  3. Apply a standard wound dressing after treatment.
  4. Apply once daily until complete debridement of necrotic tissue has been achieved. After debridement, apply the medication every other day until the wound closes (maximum treatment duration: 28 days).
  Arms: Active comparator
Drug: Placebo (Sodium Chloride Injection 0.9%) — 1. Clean the wound before applying medication.
  2. Apply Placebo (Sodium Chloride Injection 0.9%) to the wound.
  3. Apply a standard wound dressing after treatment.
  4. Apply once daily until complete debridement of necrotic tissue has been achieved. After debridement, apply the medication every other day until the wound closes (maximum treatment duration: 28 days).
  Arms: Placebo Comparator

SUMMARY:
This multicentre, randomised, double-blind, dose-finding, active- and placebo-controlled Phase II clinical trial will evaluate the safety, efficacy, pharmacokinetic profile, and immunogenicity of KJ101 for the debridement of deep second-degree burns. The trial will provide supporting evidence for subsequent Phase III trials.

DETAILED DESCRIPTION:
This multicentre, randomised, double-blind, dose-finding, active- and placebo-controlled Phase II clinical trial will evaluate the safety, efficacy, pharmacokinetic profile, and immunogenicity of KJ101 in the debridement of deep second-degree burns. The aim is to provide supporting evidence for subsequent Phase III clinical trial.

The study comprises four treatment groups: KJ101 at a dose of 800 U/mL; KJ101 at a dose of 1200 U/mL; an active comparator group receiving chymotrypsin at a dose of 800 U/mL; and a placebo control group.

Approximately 144 screened and qualified subjects will be randomised at a ratio of 1:1:1:1 to one of the four groups. All interventions will be administered locally to the target wound at the following frequencies: once daily prior to complete necrotic tissue debridement, and then every other day post-debridement.

Treatment will continue until complete wound healing is achieved (with a maximum treatment duration of 28 days), after which there will be a one-week safety follow-up period will be conducted.

ELIGIBILITY:
Inclusion criteria:

1. Male and female subjects aged 18 to 65 years inclusive, who are neither pregnant nor lactating;
2. Clinically diagnosed with superficial or deep II degree burns within 72 hours of injury, with a total burn area of ≤30% TBSA. The target burn wound must be isolated or have distinguishable boundaries, with an area between 40 and 200 cm².
3. Subjects of childbearing age must agree to use effective and safe contraceptive methods during the treatment period and for three months after the final administration.

Exclusion criteria:

1. Individuals who are known to be allergic to any component of the test drug or who have a tendency to allergies.
2. Burns caused by specific factors, such as electrical or chemical burns.
3. Subjects with shock or inhalation lung injury;
4. Subjects with target wounds complicated by inflammatory skin diseases (e.g. atopic dermatitis, eczema or psoriasis), or who have undergone enzymatic debridement (e.g. with collagenase, papain, bromelain, chymotrypsin or trypsin).
5. Subjects who, during screening, are judged by the investigator to have other severe systemic infections requiring systemic treatment;
6. Abnormal liver or kidney function.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-06-16 (Estimated); Primary Completion 2026-03-18 (Estimated); Study Completion 2026-08-29 (Estimated)

PRIMARY OUTCOMES:
Adverse events | day 35
  Assessing the incidence and severity of adverse events (AEs) and serious adverse events (SAEs) via the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

SECONDARY OUTCOMES:
The time required for burn wounds to heal completely. | day 3 to day 28
  The time taken for the burn wound to reach full epithelialisation, i.e. complete healing.
Rate of complete healing of burn wounds. | day 28
  The complete burn wound healing rate was calculated as follows:
  (Number of subjects with complete burn wound healing within 28 days of randomisation/Total number of subjects) x 100%.
  Complete wound healing of burn wounds in patients was assessed using the criterion of 100% epithelialisation of the burn wound.
The time it takes to completely remove necrotic tissue from burn wound. | day 3 to day 28
  Necrotic tissue in a wound was defined as inactive tissue that had lost its ability to heal due to irreversible cell death caused by thermal injury. The complete removal of necrotic tissue from a burn wound was defined as the point at which the wound was fully cleared of necrotic tissue, the base was clean, and new tissue had formed.
Pain intensity evaluation (VAS score) | day 1 to day 28
  A visual analogue scale (VAS) is used to assess pain. The basic method involves a 10 cm scale divided into 10 points, with '0' and '10' at each end. '0' represents no pain, while '10' represents the most severe and intolerable pain possible.
Pharmacokinetics of KJ101 (Cmax) | day 28
  Maximum observed serum concentration of KJ101 following dosing (Cmax)
Pharmacokinetics of KJ101 (AUC) | day 28
  Area under the serum concentration versustime curve (AUC)
Pharmacokinetics of KJ101 (t1/2) | day 28
  Half-life of KJ101
Pharmacokinetics of KJ101 (CL) | day 28
  Clearance(CL) is a measure of the ability of the body to clear KJ101
Pharmacokinetics of KJ101 (Vz) | day 28
  Vz = Volume of distribution during the elimination phase
Immunogenicity | day 28
  Immunogenicity of KJ101 (Anti-KJ101 antibody) in patients

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No